CLINICAL TRIAL: NCT03071068
Title: A Phase 2, Single-masked, Multicentre Study to Evaluate the Safety and Efficacy of 2 Dose Levels of THR-317 for the Treatment of Diabetic Macular Oedema (DME)
Brief Title: A Study to Evaluate the Safety and Efficacy of THR-317 for the Treatment of Diabetic Macular Oedema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THR-317-001; 2016-002100-25 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2017-03-06 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Retinopathy; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- THR-317 4mg (Experimental): anti-PlGF recombinant monoclonal antibody, 4mg dose
  Interventions: Drug: Anti-PlGF recombinant monoclonal antibody, 4mg dose
- THR-317 8mg (Experimental): anti-PlGF recombinant monoclonal antibody, 8mg dose
  Interventions: Drug: Anti-PlGF recombinant monoclonal antibody, 8mg dose

INTERVENTIONS:
Drug: Anti-PlGF recombinant monoclonal antibody, 4mg dose — 3 intravitreal injections of THR-317 4mg approximately 1 month apart
  Arms: THR-317 4mg
Drug: Anti-PlGF recombinant monoclonal antibody, 8mg dose — 3 intravitreal injections of THR-317 8mg approximately 1 month apart
  Arms: THR-317 8mg

SUMMARY:
This study is conducted to evaluate the safety of THR-317 when administered intravitreally and to assess the compound's efficacy in improving best-corrected visual acuity (BCVA) and reducing central subfield thickness (CST) in subjects with centre-involved diabetic macular oedema (DME).

ELIGIBILITY:
Inclusion criteria:

* Male or female aged 18 years or older
* Type 1 or type 2 diabetes
* Centre-involved DME with CST ≥ 340µm on Spectralis SD-OCT or ≥ 320µm on non-Spectralis SD OCT, in the study eye
* Reduced vision primarily due to DME, with BCVA between 72 and 23 ETDRS letters read at 4 meters (20/40 and 20/320 Snellen equivalent) in the study eye
* Anti-vascular endothelial growth factor (anti-VEGF) treatment naïve study eye or poor response to prior anti-VEGF treatment in the study eye
* Non-proliferative diabetic retinopathy, or stable proliferative diabetic retinopathy without neovacularisation at the disc
* Written informed consent obtained from the subject prior to screening procedures

Exclusion criteria:

* Concurrent disease in the study eye, other than DME, that could compromise BCVA, require medical or surgical intervention during the study period or could confound interpretation of the results
* Previous treatments / procedures in the study eyes as follows, or their planned use during the THR-317 treatment period for up to 30 days after the last injection: panretinal or focal / grid laser photocoagulation [3 months], anti-VEGF treatment [any time for anti-VEGF naïve subjects; 4 weeks for subjects with a poor response to anti-VEGF treatment], intra-ocular or peri-ocular corticosteroids [4 months], steroid implant [any time], intra-ocular surgery [3 months], vitrectomy [any time]
* Any active ocular / intra-ocular infection or inflammation in either eye
* Aphakic study eye
* Untreated diabetes
* Glycated haemoglobin A (HbA1c) > 12%
* Uncontrolled hypertension in the opinion of the Investigator
* Pregnant or lactating female or female of child-bearing potential not utilising an adequate form of contraception or male of reproductive potential not utilising contraception suggesting lens / zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute (up to the 7-day follow-up visit) ocular (serious) adverse events ([S]AEs) in the study eye, after each injection and across injections per subject | up to the 7-day follow-up visit after each injection

SECONDARY OUTCOMES:
Incidence of systemic and ocular (S)AEs up to the 30-day follow-up visit, after each injection and across injections per subject | up to the 30-day follow-up visit after each injection
Incidence of systemic and ocular (S)AEs from first injection up to Day 90 and up to Day 150 | From day 0 to day 150
Proportion of subjects withdrawn from repeat injection and reason for withdrawal | At day 30 and at day 60
Proportion of subjects with a loss of ≥ 15, ≥ 10 or ≥ 5 ETDRS letters in BCVA from baseline by study visit | Up to day 150
Proportion of subjects with an acute loss (up to the 7-day follow-up visit) of ≥ 15, ≥ 10 or ≥ 5 ETDRS letters in BCVA after each injection | Up to 7-day follow-up visit after each injection
Proportion of subjects with a ≥ 15 ETDRS letters gain in BCVA from baseline or ≥ 83 ETDRS letters, by study visit | Up to day 150
Mean change from baseline in BCVA, by study visit | Up to day 150
Mean change from baseline in CST, by study visit, based on spectral domain optical coherence tomography (SD-OCT), as assessed by the central reading centre (CRC) | Up to day 150

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — ThromboGenics
Locations (10):
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Slovakia (3):
  - Bratislava
  - Trenčín
  - Žilina